CLINICAL TRIAL: NCT01272661
Title: Breast for Success: A Family-Centered Intervention in Support of Breastfeeding Among High-risk Low-income Mothers in Cleveland
Brief Title: Breast for Success: A Family-Centered Intervention in Support of Breastfeeding Among High-risk Low-income Mothers
Acronym: BFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: American Academy of Pediatrics (Other); Mt. Sinai Health Care Foundation (Other)
Responsible Party: Principal Investigator, Lydia Furman, Associate Professor of Pediatrics, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: BFS-1
Record Dates: First submitted 2010-12-27; First posted 2011-01-10 (Estimated); Results first posted 2014-05-28 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Breastfeeding
Keywords: breastfeeding; low-income; high-risk; African-American; health disparity
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Enhanced Curriculum (Active Comparator): New Enhanced Breastfeeding Curriculum with 11 brief modules
  Interventions: Behavioral: Enhanced Curriculum
- Enhanced Curriculum+Breastfeeding Doula (Active Comparator): Enhanced Curriculum + mother selects a support person to learn about breastfeeding with her and support her postpartum ("breastfeeding doula")
  Interventions: Behavioral: Enhanced Curriculum+Breastfeeding Doula
- Enhanced Curriculum +Father Support (Active Comparator): Enhanced Curriculum+ mother provides father-friendly information about breastfeeding to her partner plus an invitation to an educational group for fathers
  Interventions: Behavioral: Enhanced Curriculum +Father Support

INTERVENTIONS:
Behavioral: Enhanced Curriculum — Brief health literacy focused modules on breastfeeding delivered in the home by Community Health Workers
  Arms: Enhanced Curriculum
Behavioral: Enhanced Curriculum+Breastfeeding Doula — In the Doula Program, the Community Health Worker and mother will identify a support person (e.g. grandma, father, friend) who commits to learning about breastfeeding with the mother at home visits, and then helps her with breastfeeding postpartum.
  Arms: Enhanced Curriculum+Breastfeeding Doula
Behavioral: Enhanced Curriculum +Father Support — In the Father Support Program, mothers will give their partners father-friendly breastfeeding information and an invitation to a 3-week breastfeeding education group for fathers that includes a resource specialist or resource information for child support, re-entry and job services.
  Arms: Enhanced Curriculum +Father Support

SUMMARY:
Breast for Success is a new direct service program focused on overcoming barriers to breastfeeding for low-income inner-city mothers by use of a culturally competent and home-based educational and support intervention. Key project components include a new Enhanced Breastfeeding Curriculum with brief engaging health literacy focused modules, and two innovative support plans, the Breastfeeding Doula and Father Support Programs. The objective is to increase breastfeeding rates for high-risk inner-city mothers.

Research Questions to evaluate project feasibility and effectiveness are:

1. Were all aspects of the Curriculum and Doula and Father Support Programs implemented?
2. Is there an increase in the rate of any breastfeeding at 1 month postpartum for all mothers?
3. Is there a difference in the rate of any breastfeeding at 1 month postpartum between interventions (Curriculum only, Curriculum+Doula Support, Curriculum+Father Support)?
4. What are exclusive breastfeeding rates at 1, 3 and 6 months for all mothers?

DETAILED DESCRIPTION:
Low rates of breastfeeding among low-income inner-city mothers represent a challenging health disparity that adversely impacts child and maternal health. The overall objective of Breast for Success is to increase the rates of breastfeeding initiation, continuation and exclusivity among high-risk mothers in the City of Cleveland via home-based culturally appropriate interventions. Key project components include a new Curriculum with brief engaging modules utilizing games, teach-reteach strategies, and interactive learning to address specific barriers identified in focus groups (e.g. pain, low milk supply, breast "myths"), and two innovative support components, the Breastfeeding Doula and Father Support Programs. Breast for Success was developed in collaboration with and will be disseminated in partnership with the Cleveland Department of Public Health MomsFirst initiative (a Healthy Start Program), which delivers comprehensive services including twice-monthly Community Health Worker home visits prenatally through 2 years postpartum to 500 women annually. The investigators will measure program success via participation logs, satisfaction questionnaires and breastfeeding rates at 1, 3 and 6 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman enrolled in MomsFirst Program of Greater Cleveland

Exclusion Criteria:

* incarceration

Other study populations include the Community Health Workers, the doulas and the fathers of the study mothers.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1296 (Actual)
Dates: Start 2011-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lydia M Furman, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- MomsFirst, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Curriculum +Father Support: Enhanced Curriculum+ mother provides father-friendly information about breastfeeding to her partner plus an invitation to an educational group for fathers
  Enhanced Curriculum+Father Support Program: In the Father Support Program, mothers will give their partners father-friendly breastfeeding information and an invitation to a 3-week breastfeeding education group for fathers that includes a resource specialist or resource information for child support, re-entry and job services.
Period: Overall Study
Arm/Group | Enhanced Curriculum | Enhanced Curriculum+Breastfeeding Doula | Enhanced Curriculum +Father Support
Started | 413 | 497 | 386
Completed | 287 | 288 | 314
Not Completed | 126 | 209 | 72
Not completed — lost to followup/case closed/ no birth | 126 | 209 | 72

BASELINE CHARACTERISTICS:
Groups:
- Enhanced Curriculum+Father Support: Enhanced Curriculum+ mother provides father-friendly information about breastfeeding to her partner plus an invitation to an educational group for fathers
  Enhanced Curriculum+Father Support Program: In the Father Support Program, mothers will give their partners father-friendly breastfeeding information and an invitation to a 3-week breastfeeding education group for fathers that includes a resource specialist or resource information for child support, re-entry and job services.
- Total: Total of all reporting groups
Arm/Group | Enhanced Curriculum | Enhanced Curriculum+Breastfeeding Doula | Enhanced Curriculum+Father Support | Total
Number analyzed (Participants) | 413 | 497 | 386 | 1296
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.2 (4.8) | 22.2 (4.4) | 23.1 (4.9) | 22.2 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 413 | 497 | 386 | 1296
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 413 | 497 | 386 | 1296

OUTCOME MEASURES:

1. Primary Outcome: Program Feasibility- Feeding Outcome Collected
Description: Measure program feasibility by number of participants who were exposed to the intervention for whom there is any feeding outcome
Time Frame: by 24 months
Population: Total number of eligible MomsFirst participants who agreed to data sharing. Outcome shows number w/ any feeding outcome (not lost to follow up, no live birth, case closed by MomsFirst). This is for a 24 month period since all data was de-identified and stripped of dates so unable to specify for 12 month period
Measure: Number; unit: participants
Groups:
- Enhanced Curriculum+Father Support Program: Enhanced Curriculum+ mother provides father-friendly information about breastfeeding to her partner plus an invitation to an educational group for fathers
  Enhanced Curriculum+Father Support Program: In the Father Support Program, mothers will give their partners father-friendly breastfeeding information and an invitation to a 3-week breastfeeding education group for fathers that includes a resource specialist or resource information for child support, re-entry and job services.
Arm/Group | Enhanced Curriculum | Enhanced Curriculum+Breastfeeding Doula | Enhanced Curriculum+Father Support Program
Number analyzed (Participants) | 413 | 497 | 386
participants | 287 | 288 | 314

2. Primary Outcome: Program Feasibility - Curriculum Modules
Description: Measure program feasibility by counting the number of Breastfeeding Curricular modules that were presented of total possible = 11
Time Frame: by 24 months from program start
Measure: Mean (Inter-Quartile Range); unit: modules presented
Arm/Group | Enhanced Curriculum | Enhanced Curriculum+Breastfeeding Doula | Enhanced Curriculum+Father Support Program
Number analyzed (Participants) | 287 | 288 | 314
modules presented | 4 [1 to 7] | 3 [0 to 6] | 2 [0 to 6]

3. Secondary Outcome: Breastfeeding Rate
Description: Measure rate of any breastfeeding (breastfeeding initiation) in the hospital. We will also compare this rate between the 3 intervention groups.
Time Frame: Any breastfeeding: participants were followed for the duration of hospital stay, an average of 48 hours
Population: ITT analysis was conducted on participants with available data
Measure: Number; unit: participants
Arm/Group | Enhanced Curriculum | Enhanced Curriculum+Breastfeeding Doula | Enhanced Curriculum+Father Support Program
Number analyzed (Participants) | 99 | 122 | 194
participants | 66 | 98 | 152

4. Secondary Outcome: Breastfeeding Rate at One Month Postpartum
Description: Measure rate of breastfeeding (rate of any breastfeeding is main measure, also measure rate of exclusive breastfeeding) at one month postpartum. Will compare rate of any breastfeeding one month postpartum to historical data, and will compare rates of any breastfeeding at one month postpartum between intervention groups.
Time Frame: Any and exclusive breastfeeding at one month, between 21-38 days postpartum
Population: ITT analysis conducted on participants with available data
Measure: Number; unit: participants
Arm/Group | Enhanced Curriculum | Enhanced Curriculum+Breastfeeding Doula | Enhanced Curriculum+Father Support Program
Number analyzed (Participants) | 243 | 222 | 259
participants | 100 | 95 | 134

5. Secondary Outcome: Breastfeeding Rate at 3 Months Postpartum
Description: Measure rates of any and exclusive breastfeeding at 3 months postpartum. Rate of any breastfeeding is presented.
Time Frame: Any and exclusive breastfeeding at 3 months, between 10-14 weeks postpartum
Population: ITT analysis conducted on participants with available data
Measure: Number; unit: participants
Arm/Group | Enhanced Curriculum | Enhanced Curriculum+Breastfeeding Doula | Enhanced Curriculum+Father Support Program
Number analyzed (Participants) | 184 | 189 | 262
participants | 48 | 44 | 67

6. Secondary Outcome: Breastfeeding Rate at 6 Months Postpartum
Description: Measure breastfeeding rate (any and exclusive) at 6 months postpartum. Rate of any breastfeeding is presented.
Time Frame: Any and exclusive breastfeeding at 6 months, between 22-26 weeks postpartum
Population: ITT analysis conducted on participants with available data
Measure: Number; unit: participants
Arm/Group | Enhanced Curriculum | Enhanced Curriculum+Breastfeeding Doula | Enhanced Curriculum+Father Support Program
Number analyzed (Participants) | 148 | 127 | 237
participants | 22 | 18 | 38

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events were not identified.
Arm/Group | Enhanced Curriculum | Enhanced Curriculum+Breastfeeding Doula | Enhanced Curriculum+Father Support Program
Serious Adverse Events (participants affected / at risk) | 0/413 | 0/497 | 0/386
Other Adverse Events (participants affected / at risk) | 0/413 | 0/497 | 0/386

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No